CLINICAL TRIAL: NCT01739270
Title: Dexamethasone Added to Levobupivacaine Improves Postoperative Analgesia After Supraclavicular Brachial Plexus Blockade
Brief Title: Dexamethasone Added to Levobupivacaine Improves Postoperative Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Jasminka Persec, MD, PhD, Anesthesiology, Resuscitation and Intensive Care Medicine Specialist, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0911
Record Dates: First submitted 2012-11-25; First posted 2012-12-03 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Brachial Plexus Anesthesia; Analgesia
Keywords: analgesia; regional anesthesia; surgery; duration of analgesia; dexamethasone added to levobupivacaine compared to levobupivacaine alone
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexamethasone with levobupivacaine (Active Comparator): 25ml 0.5% levobupivacaine plus 4mg Dexamethasone are given for supraclavicular brachial plexus block for upper extremity surgery
  Interventions: Procedure: supraclavicular brachial plexus block
- levobupivacaine (Active Comparator): 25ml 0.5% levobupivacaine plus 1ml 0.9% saline are given for supraclavicular brachial plexus block for upper extremity surgery
  Interventions: Procedure: supraclavicular brachial plexus block

INTERVENTIONS:
Procedure: supraclavicular brachial plexus block

SUMMARY:
Adding dexamethasone to local anesthetic will significantly prolong duration of brachial plexus anesthesia and analgesia.

DETAILED DESCRIPTION:
Operations of upper extremities are often performed in regional anesthesia blocks. Single-injection blocks are effective, but time limited. Adding 4mg of dexamethasone to 0.5% levobupivacaine will significantly prolong duration of brachial plexus anesthesia and analgesia for fracture operations of upper extremity. This effect will result in less opioid use postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or older
* ASA (American Society of Anesthesiologists) physical status I, II or III

Exclusion Criteria:

* refusal of the patients to give informed consent
* preexisting coagulation disorders
* local infection at the site of the block
* neuropathy
* drug or alcohol abusers
* known allergy to the drug used in study
* operation time exceeding six hours

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
duration of analgesia | 24 hour postoperatively
  Duration of analgesia after supraclavicular block

SECONDARY OUTCOMES:
postoperative analgesic consumption | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Ino Husedzinovic, Professor, Study Chair — Clinical Hospital Dubrava, Head of Anesthesiology, Resuscitation and Intensive Care Medicine
Locations (1):
- Clinical Hospital Dubrava, Zagreb, Croatia

REFERENCES:
- [Result] Parrington SJ, O'Donnell D, Chan VW, Brown-Shreves D, Subramanyam R, Qu M, Brull R. Dexamethasone added to mepivacaine prolongs the duration of analgesia after supraclavicular brachial plexus blockade. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):422-6. doi: 10.1097/AAP.0b013e3181e85eb9. PMID 20814282
- [Result] Vieira PA, Pulai I, Tsao GC, Manikantan P, Keller B, Connelly NR. Dexamethasone with bupivacaine increases duration of analgesia in ultrasound-guided interscalene brachial plexus blockade. Eur J Anaesthesiol. 2010 Mar;27(3):285-8. doi: 10.1097/EJA.0b013e3283350c38. PMID 20009936
- [Result] Kim YJ, Lee GY, Kim DY, Kim CH, Baik HJ, Heo S. Dexamathasone added to levobupivacaine improves postoperative analgesia in ultrasound guided interscalene brachial plexus blockade for arthroscopic shoulder surgery. Korean J Anesthesiol. 2012 Feb;62(2):130-4. doi: 10.4097/kjae.2012.62.2.130. Epub 2012 Feb 20. PMID 22379567